CLINICAL TRIAL: NCT04969926
Title: Natural History Study of Parathyroid Disorders
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000344; 000344-DK
Record Dates: First submitted 2021-07-20; First posted 2021-07-21 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11-21

CONDITIONS: Parathyroid Cancer; Primary Hyperparathyroidism; Pseudohypoparathyroidism; Inheritable Bone Diseases; Multiple Endocrine Neoplasia, Type 1
Keywords: Hyperparathyroidism; calcium disorders; Parathyroid Cancer; Inheritable; PSEUDOHYPOPARATHYROIDISM; Natural History
MeSH Terms: conditions — Parathyroid Neoplasms; Hyperparathyroidism, Primary; Pseudohypoparathyroidism; Multiple Endocrine Neoplasia Type 1; Hyperparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with confirmed, suspected or at risk of developing parathyroid disorder: Parathyroid (and related disorders) will be evaluated and their biospecimens collected to define the molecular signature and clinical spectrum of their disorder

SUMMARY:
Background:

Parathyroid disorders are very common in the general population and include disorders of parathyroid excess, deficiency, or defects in parathyroid hormone (PTH) signaling. PTH, the main secretory product of parathyroid glands is responsible for regulation of calcium-phosphate homeostasis.

Objective:

i) To investigate the cause of parathyroid disorders

ii) To describe evolution, natural history, and longitudinal trends of parathyroid and related disorders seen in syndromic presentations like multiple endocrine neoplasia, hyperparathyroidism-jaw tumor syndrome

Eligibility:

People ages 6 months older who have, are at risk of having, or are related to a person with a parathyroid or related disorder.

Design:

Participants will be screened with a review of their medical records.

Participants will be seen, tested, and treated by doctors based on their condition. Their visits may be in person or via telehealth.

Participants will complete questionnaires. They will answer questions about their physical, mental, and social health.

Participants may give samples such as saliva, blood, urine, or stool.

Participants may give cheek cell samples. They will do this using a cheek swab or by spitting into a cup.

Adult participants may give a skin biopsy. For this, a small bit of skin is removed with a punch tool.

Participants may have medical photos taken.

If participants have surgery during the course of their regular care either at the NIH

or at a different hospital or doctor s office, researchers will ask for some of the leftover

tissue.

Participants will be in the study as long as they are being seen by their doctor.

DETAILED DESCRIPTION:
Study Description:

Patients with confirmed, suspected or at risk of developing parathyroid disorders will be provided standard of care testing for their condition. Data obtained during the testing will be used for research. Additionally, samples may be collected for research.

Objectives:

* To investigate the cause of the disease and its associated manifestations, possibly genetic in participants with parathyroid and related disorder(s)
* To identify biomarkers of the various parathyroid disorder(s) and associated manifestations by performing molecular profiling of available biospecimens
* To describe evolution, natural history and longitudinal trends of parathyroid and related disorders including the associated extra- parathyroid manifestations seen in these disorders, for example, Zollinger-Ellison syndrome, gastro-entero-pancreatic neuroendocrine tumors, kidney, jaw, pituitary and uterine tumors.
* To investigate the natural history of parathyroid disorders and associated manifestations during pregnancy
* To characterize the morbidity and mortality in participants with parathyroid and related disorders and investigate its association with extra-parathyroidal manifestations.
* To investigate long-term risks and benefits with standard of care testing and therapy for parathyroid and associated extra-parathyroidal manifestations.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Subjects known to have, suspected of having, or at risk of developing a parathyroid or related disorder.
* Age >= 6 months.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Children <= 6 months
* Patients with conditions that in the opinion of the investigators can interfere with the study objectives.

Ages: 6 Months to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with confirmed, suspected or at risk of developing parathyroid and related disorders.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2031-01-22 (Estimated); Study Completion 2031-01-22 (Estimated)

PRIMARY OUTCOMES:
To identify biomarkers of the disease and associated manifestations by performing molecular profiling of available biospecimens | 5 years
  Participants will undergo standard clinical evaluations for their condition. Data obtained during these evaluations will be retained for purposes of the primary objective, for analysis of secondary objectives, and for future research. There are no mandatory study procedures for this protocol.
To investigate the cause and molecular mechanism of the disease, possibly genetic in participants with unknown cause of parathyroid and related disorder(s) | 5 years
  Participants will undergo standard clinical evaluations for their condition. Data obtained during these evaluations will be retained for purposes of the primary objective, for analysis of secondary objectives, and for future research. There are no mandatory study procedures for this protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Smita Jha, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Worthy CC, Tora R, Uttarkar CN, Welch JM, Bliss L, Cochran C, Ninan A, Kumar S, Wank S, Auh S, Weinstein LS, Simonds WF, Agarwal SK, Blau JE, Jha S. Genotype-phenotype correlation in multiple endocrine neoplasia type 1. JCI Insight. 2025 Feb 13;10(6):e176993. doi: 10.1172/jci.insight.176993. PMID 39946193
- [Derived] Graf A, Cochran C, Sadowski S, Nilubol N, Simonds WF, Weinstein LS, Chang R, Jha S. Invasive Testing for Preoperative Localization of Parathyroid Tumors. J Endocr Soc. 2024 Jan 2;8(1):bvad158. doi: 10.1210/jendso/bvad158. eCollection 2023 Dec 1. PMID 38174154
- [Derived] Tora R, Welch J, Sun J, Agarwal SK, Bell DA, Merino M, Weinstein LS, Simonds WF, Jha S. Phenotypic Profiling and Molecular Mechanisms in Hyperparathyroidism-jaw Tumor Syndrome. J Clin Endocrinol Metab. 2023 Nov 17;108(12):3165-3177. doi: 10.1210/clinem/dgad368. PMID 37339334
- [Derived] Zenno A, Ramamoorthy B, Hammoud DA, Quezado M, Zeiger MA, Jha S. Case Report: Nine-year-old with parathyroid adenoma within the piriform sinus. Front Endocrinol (Lausanne). 2023 May 23;14:1171052. doi: 10.3389/fendo.2023.1171052. eCollection 2023. PMID 37288292
- [Derived] Chuki E, Graf A, Ninan A, Tora R, Abijo T, Bliss L, Nilubol N, Weinstein LS, Agarwal SK, Simonds WF, Jha S. Long-Term Outcomes of Parathyroid Autografts in Primary Hyperparathyroidism. J Endocr Soc. 2023 Apr 22;7(5):bvad055. doi: 10.1210/jendso/bvad055. eCollection 2023 Mar 6. PMID 37284613
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000344-DK.html